CLINICAL TRIAL: NCT02567409
Title: A Randomized Phase 2 Trial of Cisplatin/Gemcitabine With or Without M6620 (VX-970) in Metastatic Urothelial Carcinoma
Brief Title: Cisplatin and Gemcitabine Hydrochloride With or Without Berzosertib in Treating Patients With Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01642; NCI-2015-01642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-135; 9947 (Other: City of Hope Comprehensive Cancer Center LAO); 9947 (Other: CTEP); N01CM00038 (NIH); UM1CA186690 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis and Ureter Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Stage IV Bladder Urothelial Carcinoma AJCC v7
MeSH Terms: interventions — berzosertib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (berzosertib, gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and cisplatin IV over 60 minutes on day 1. Patients also receive berzosertib IV over 60 minutes on days 2 and 9. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berzosertib; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride
- Arm B (gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive gemcitabine hydrochloride and cisplatin as in Arm A.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
  Arms: Arm A (berzosertib, gemcitabine hydrochloride, cisplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011

SUMMARY:
This phase II trial studies how well cisplatin and gemcitabine hydrochloride with or without berzosertib works in treating patients with urothelial cancer that has spread to other places in the body (metastatic). Drugs used in chemotherapy, such as cisplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Berzosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known if cisplatin and gemcitabine hydrochloride work better alone or with berzosertib in treating patients with urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the addition of berzosertib (M6620 [VX-970]) to cisplatin/gemcitabine hydrochloride (gemcitabine) improves progression-free survival (PFS) relative to cisplatin/gemcitabine alone.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) with the addition of M6620 (VX-970) to cisplatin/gemcitabine relative to cisplatin/gemcitabine alone.

II. To compare tumor response rate with the addition of M6620 (VX-970) to cisplatin/gemcitabine relative to cisplatin/gemcitabine alone.

III. To compare safety with the addition of M6620 (VX-970) to cisplatin/gemcitabine relative to cisplatin/gemcitabine alone.

IV. To assess the role of p53 status in predicting response to M6620 (VX-970)-based therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8, and cisplatin IV over 60 minutes on day 1. Patients also receive berzosertib IV over 60 minutes on days 2 and 9. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive gemcitabine hydrochloride and cisplatin as in Arm A.

After completion of study treatment, patients are followed up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic urothelial carcinoma; urothelial cancer derived from the bladder, ureter or upper tract is permitted
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have access to archival tumor tissue for proposed correlative studies; these may be derived from transurethral resection of bladder tumors (TURBT), cystectomy, or biopsy; if archival tissue is not available for proposed correlatives, patients may be enrolled at the discretion of the study principal investigator (PI) (SKP)
* No prior cytotoxic chemotherapy for metastatic disease; prior immunotherapy is permitted
* At least 12 months have elapsed since platinum-based peri-operative treatment
* Karnofsky >= 70% (Eastern Cooperative Oncology Group [ECOG] performance status 0-1)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine clearance >= 50 mL/min by either measured (using the Cockcroft-Gault, Modification of Diet in Renal Disease [MDRD] or Chronic Kidney Disease Epidemiology [CKD-EPI] formula) or calculated clearance (i.e. glomerular filtration rate [GFR])
* The effects of M6620 (VX-970) on the developing human fetus are unknown; for this reason and because DNA-damage response (DDR) inhibitors as well as other therapeutic agents used in this trial may have teratogenic potential, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of M6620 (VX-970) administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Radiotherapy within 4 weeks of protocol therapy
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX970), cisplatin, or gemcitabine
* M6620 (VX-970) is primarily metabolized by CYP3A4; therefore, concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of; Patient Drug Information Handout and Wallet Card should be provided to patients; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because M6620 (VX-970) as a DNA-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970), breastfeeding should be discontinued if the mother is treated with M6620 (VX-970); these potential risks may also apply to other agents used in this study
* Patients with >= grade 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (39):
- United States (39):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Pal SK, Frankel PH, Mortazavi A, Milowsky M, Vaishampayan U, Parikh M, Lyou Y, Weng P, Parikh R, Teply B, Dreicer R, Emamekhoo H, Michaelson D, Hoimes C, Zhang T, Srinivas S, Kim WY, Cui Y, Newman E, Lara PN Jr. Effect of Cisplatin and Gemcitabine With or Without Berzosertib in Patients With Advanced Urothelial Carcinoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1536-1543. doi: 10.1001/jamaoncol.2021.3441. PMID 34436521

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin): Patients receive cisplatin, 60 mg/m2, on day 1; gemcitabine, 875 mg/m2, on days 1 and 8; and berzosertib, 90 mg/m2, on days 2 and 9 of a 21-day cycle.
  Berzosertib: Given IV
  Cisplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
- Arm B (Gemcitabine Hydrochloride, Cisplatin): Patients receive cisplatin,70 mg/m2, on day 1 and gemcitabine, 1000 mg/m2, on days 1 and 8 of a 21-day cycle
  Cisplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
Started | 46 | 41
Completed | 46 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin) | Total
Number analyzed (Participants) | 46 | 41 | 87
Age, Continuous [Median (Full Range); unit: years] | 67.5 [32 to 82] | 65 [32 to 84] | 66 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 38 | 30 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 1 | 2
  White Not Hispanic | 38 | 34 | 72
  Asian | 2 | 1 | 3
  African American | 4 | 3 | 7
  Unknown | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 46 | 41 | 87
Prior Neoadjuvant Cisplatin [Count of Participants; unit: Participants]
  Yes | 5 | 4 | 9
  No | 41 | 37 | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Day of randomization, until progression, or death, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
Number analyzed (Participants) | 46 | 41
Months | 8.0 [6.0 to 14.4] | 8.0 [6.8 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) vs Arm B (Gemcitabine Hydrochloride, Cisplatin); Test type: Superiority; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.69 to 1.98] — Hazard ratio relative to arm B

2. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as death from any cause.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
Number analyzed (Participants) | 46 | 41
Months | 14.4 [10.0 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 19.8 [14.8 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) vs Arm B (Gemcitabine Hydrochloride, Cisplatin); Test type: Superiority; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.71 to 2.48] — Hazard ratio relative to arm B

3. Secondary Outcome: Confirmed Objective Response Rate
Description: Response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Confirmed Objective Response = CR + PR.
Time Frame: Up to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
Number analyzed (Participants) | 46 | 41
percentage of participants | 54 [39 to 69] | 63 [47 to 78]
Statistical Analysis 1: Comparison: Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) vs Arm B (Gemcitabine Hydrochloride, Cisplatin); Test type: Superiority; p = 0.51, Fisher Exact

4. Secondary Outcome: Treatment Limiting Adverse Events
Description: Adverse events that were fatal or led to treatment discontinuation.
Time Frame: Assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
Number analyzed (Participants) | 46 | 41
Participants
  Hypotension | 0 | 1
  Multi-organ failure | 0 | 1
  Cardiac arrest | 1 | 0
  Neutropenia | 2 | 0
  Respiratory failure | 1 | 0
  Pulmonary embolism | 1 | 1
  Thrombocytopenia | 2 | 2
  Creatinine Increased | 1 | 2
  Leukocytosis | 1 | 0
  Acute kidney injury | 1 | 0
  Vomiting | 0 | 1
  Urinary tract infection | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 36 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) | Arm B (Gemcitabine Hydrochloride, Cisplatin)
All-Cause Mortality (participants affected / at risk) | 29/46 | 25/41
Serious Adverse Events (participants affected / at risk) | 29/46 | 12/41
Other Adverse Events (participants affected / at risk) | 40/46 | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) (N=46) | Arm B (Gemcitabine Hydrochloride, Cisplatin) (N=41)
Anemia (Blood and lymphatic system disorders) | 14 (23) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Edema limbs (General disorders) | 2 (2) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (7) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (11) | 0 (0)
Platelet count decreased (Investigations) | 15 (28) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 6 (9) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Disease progression (General disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 0 (0)
Nephrostomy Tube Malfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (6) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (7)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
prostatic abscess (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 2 (3)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Berzosertib, Gemcitabine Hydrochloride, Cisplatin) (N=46) | Arm B (Gemcitabine Hydrochloride, Cisplatin) (N=41)
Anemia (Blood and lymphatic system disorders) | 36 (262) | 26 (193)
Blood LDH Increased (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Blood LDH increased (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased WBC count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left groin mass oozing (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
WBC count increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
thrombocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (6) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (3)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 6 (18) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 4 (5)
Tinnitus (Ear and labyrinth disorders) | 4 (13) | 5 (17)
Blurred vision (Eye disorders) | 1 (1) | 2 (3)
Right eye vision (Eye disorders) | 0 (0) | 1 (2)
Visual acuity decreased (Eye disorders) | 1 (1) | 0 (0)
right eye vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (13) | 7 (21)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (32) | 16 (47)
Diarrhea (Gastrointestinal disorders) | 11 (20) | 9 (18)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 2 (8)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gas pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 6 (18)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mouth Sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (5)
Nausea (Gastrointestinal disorders) | 29 (101) | 23 (104)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sore tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (5) | 0 (0)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (25) | 15 (31)
hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
indegestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (4)
Chattering teeth without chills (General disorders) | 0 (0) | 1 (5)
Chills (General disorders) | 6 (8) | 2 (3)
Edema face (General disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 11 (37) | 6 (21)
Fatigue (General disorders) | 26 (114) | 26 (121)
Fever (General disorders) | 11 (15) | 4 (10)
Flu like symptoms (General disorders) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 2 (7) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Hypoproteinemia (General disorders) | 4 (5) | 3 (7)
Hyporteinemia (General disorders) | 1 (1) | 0 (0)
Increased Blood Urea (General disorders) | 2 (2) | 1 (1)
IncreasedBlood urea (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 6 (6) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 3 (4)
Injection site reaction (General disorders) | 3 (5) | 2 (5)
LDH level (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (6) | 0 (0)
Lump to back of neck (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (5) | 1 (3)
Pain (General disorders) | 8 (14) | 2 (2)
Raised Blood Urea (General disorders) | 1 (1) | 0 (0)
Redness around Infusion site (General disorders) | 1 (1) | 0 (0)
Right Nipple Sensation Intermittent (General disorders) | 1 (2) | 0 (0)
Weakness (General disorders) | 0 (0) | 1 (1)
diaphoresis (General disorders) | 1 (1) | 0 (0)
edema of limb (General disorders) | 0 (0) | 1 (1)
functional status decline (General disorders) | 0 (0) | 1 (1)
pain at infusion site (General disorders) | 0 (0) | 1 (1)
pain at portal site (General disorders) | 0 (0) | 1 (1)
right nipple sensation intermittent (General disorders) | 1 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (3) | 0 (0)
cold sores (Immune system disorders) | 1 (1) | 0 (0)
Cold Symptoms (Infections and infestations) | 0 (0) | 1 (3)
Cold symptoms (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 1 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Leaking left inguinal area from tumor si (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (2)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis of unknown origin (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Skin infection (Infections and infestations) | 3 (4) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (9) | 6 (10)
ear infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 5 (10) | 2 (4)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cut on Finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Tear (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
firmness of vein in left arm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
firmness of vein in right arm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
firmness, swelling of vein on back of ri (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
firmness/swelling of vein on back of rig (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
knot in left arm distal to elbow (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
AST, decreased (Investigations) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 8 (16) | 9 (19)
Alkaline phosphatase increased (Investigations) | 12 (39) | 13 (48)
Aspartate aminotransferase increased (Investigations) | 9 (20) | 8 (21)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (7) | 1 (1)
Blood Lactate Dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (8) | 2 (10)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (2) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 19 (67) | 17 (83)
Glucosuria (Investigations) | 0 (0) | 1 (4)
Hyperphosphatemia (Investigations) | 3 (5) | 3 (5)
Increased Blood urea (Investigations) | 1 (1) | 2 (2)
Increased LDH (Investigations) | 0 (0) | 1 (1)
Increased Lactic Dehdrogenase (Investigations) | 1 (1) | 0 (0)
IncreasedLDH (Investigations) | 0 (0) | 1 (1)
IncreasedPhosphate (Investigations) | 1 (1) | 0 (0)
Inreased LDH (Investigations) | 0 (0) | 1 (1)
LDH increased (Investigations) | 4 (17) | 2 (4)
Lactate Dehydrogenase Increased (Investigations) | 1 (6) | 0 (0)
Lactic acid increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 14 (94) | 14 (60)
Neutrophil count decreased (Investigations) | 23 (78) | 20 (55)
Phosphorus Increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 34 (212) | 23 (162)
Procalcitonin, increased (Investigations) | 1 (1) | 0 (0)
Reduced Bicarbonate (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 2 (5) | 1 (2)
Weight loss (Investigations) | 8 (21) | 7 (29)
White blood cell decreased (Investigations) | 19 (88) | 15 (56)
hyperphosphatemia (Investigations) | 1 (1) | 0 (0)
hypoproteinemia (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 11 (31) | 10 (44)
DECREASED ALT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DECREASED AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (10) | 7 (8)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (28) | 11 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (13) | 6 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (49) | 10 (39)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (23) | 14 (38)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 10 (35) | 11 (40)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (28) | 10 (30)
Hyponatremia (Metabolism and nutrition disorders) | 21 (59) | 20 (59)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (21) | 10 (21)
Increased ALT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased AST (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Raised LDH (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (21) | 6 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (15) | 1 (6)
Calf tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (20) | 6 (10)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (10) | 4 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 6 (14)
Pulled muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Umbiliclal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Altered Mental status (Nervous system disorders) | 1 (1) | 0 (0)
Disorientation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (21) | 10 (15)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (27) | 6 (22)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 5 (23) | 7 (23)
Paresthesia (Nervous system disorders) | 7 (12) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (8) | 5 (11)
Presyncope (Nervous system disorders) | 2 (2) | 2 (3)
Stroke (Nervous system disorders) | 0 (0) | 1 (3)
Tremor (Nervous system disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (7) | 2 (4)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (9) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (20) | 5 (17)
Vivid dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 3 (11)
Bladder spasm (Renal and urinary disorders) | 1 (2) | 1 (5)
Chronic kidney disease (Renal and urinary disorders) | 4 (9) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (20) | 4 (8)
Hydronephrosis (Renal and urinary disorders) | 3 (5) | 2 (2)
Neph Tube not draining (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrostomy tube malfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (16) | 4 (12)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (5)
Urinary incontinence (Renal and urinary disorders) | 1 (4) | 1 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 1 (3)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BILATERAL LOWER LUNG RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 4 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (20) | 5 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (8)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 5 (17)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 3 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (9)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
dry mucus membranes with blood mixed int (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Callus (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Facial Petechia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Melanoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (3)
RIGHT WRIST ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Rash NOS (Leg Petechia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (8)
Rash over back and abdomen (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3)
Tenderness left upper arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Tinea crusis (groin) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
tinea cruris (groin) (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Mediport Placement (Surgical and medical procedures) | 1 (1) | 0 (0)
DVT (Vascular disorders) | 0 (0) | 1 (4)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 10 (31) | 9 (32)
Hypotension (Vascular disorders) | 7 (10) | 1 (1)
Peripheral artery disease (Vascular disorders) | 0 (0) | 1 (4)
Petechiae (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 5 (9) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 6 (13) | 5 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT02567409/Prot_SAP_000.pdf